CLINICAL TRIAL: NCT01974739
Title: Hypernatraemia and Diuretics in Intensive Care Patients
Brief Title: Hydrochloorthiazide and Hypernatriaemie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, E.C. Boerma, MD PhD, Frisius Medisch Centrum
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABR 44878
Record Dates: First submitted 2013-10-28; First posted 2013-11-04 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Hypernatraemia
Keywords: intensive care; diuretics
MeSH Terms: conditions — Hypernatremia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- hydrochloorthiazide (Active Comparator): once a day 25 mg
  Interventions: Drug: Hydrochloorthiazide
- placebo (Placebo Comparator): once a day placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Hydrochloorthiazide
  Arms: hydrochloorthiazide
Drug: placebo
  Arms: placebo

SUMMARY:
Acquired hypernatremia appears to be associated with mortallity in ICU. To reduce hypernatremia and shorten the time of hypernatremia, we investigate the effect of hydrochloorthiazide compared to a placebo

ELIGIBILITY:
Inclusion Criteria:

* sodium > 142

Exclusion Criteria:

* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
sodium level | 7 days
  a decrease of 5 mmol/L sodium in plama

SECONDARY OUTCOMES:
time hypernatraemia | 7 days
  decrease of duration high sodium level in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Christiaan Boerma, MD, Principal Investigator — Frisius Medisch Centrum
Locations (1):
- Medical Centre Leeuwarden, Leeuwarden, Provincie Friesland, Netherlands